CLINICAL TRIAL: NCT05451017
Title: The Effect of Food on the Oral Bioavailability of AEF0117 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was initially paused due to a research hold of the institution. However, the study will not continue as the sample size of patients collected prior to the pause allowed for adequate data analysis of the study endpoints.
Sponsor: Aelis Farma (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AEF0117-105; U01DA053832 (NIH)
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Marijuana Abuse
Keywords: AEF0117; Cannabis-related Use Disorder; Cannabis subjective effects; Cannabis self-administration cannabis-induced analgesia; Cannabis-related cognitive disorder
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, parallel-group, 2-arm, open-label, single-dose trial in healthy male and female volunteers aged 18-55 years to obtain data on the effect of food on the oral bioavailability of AEF0117.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AEF0117 1.0 mg in fasted condition (Experimental): 16 participants receive 1 dose of AEF0117 1 mg in fasted condition
  Interventions: Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one in fasting condition
- AEF0117 1.0 mg in fed condition (Experimental): 16 participants receive 1 dose of AEF0117 1 mg fed condition
  Interventions: Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one in fed condition

INTERVENTIONS:
Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one in fed condition — a single dose of 1 mg AEF0117 in fed condition
  Other Names: AEF0117
  Arms: AEF0117 1.0 mg in fed condition
Drug: 3ß-(4-methoxybenzyloxy)pregn-5-en-20-one in fasting condition — a single dose of 1 mg AEF0117 in fasting condition
  Other Names: AEF0117
  Arms: AEF0117 1.0 mg in fasted condition

SUMMARY:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders.

In the 3 early studies conducted with AEF0117, AEF0117 was administered orally after a light breakfast. AEF0117 showed a good bioavailability and favorable, dose-proportional pharmacokinetics . In this protocol, the effects of food on AEF0117 bioavailability in healthy volunteers will be investigated by comparing the rate and extent of AEF0117 when 1 mg AEF0117 is administered in fed state versus fasting state.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date. This trial will provide data on the effect of food on the oral bioavailability of AEF0117 to support the next stage of the clinical development of the drug.

DETAILED DESCRIPTION:
Cannabis is the most widely used illicit drug with approximately 28 million individuals reporting past-month use, and 14% of those receiving substance use disorder treatment in the US reporting cannabis as their primary drug of abuse. While psychotherapeutic approaches have some utility for treating Cannabis Use Disorder (CUD), the vast majority of patients have difficulty significantly reducing their use or achieving abstinence. Safe and effective medications to treat CUD are urgently needed. The overall goal of this clinical trial is to contribute to advancing a safe and effective pharmacotherapy for CUD along the FDA approval pipeline.

When the CB1 receptors are over-activated by very high doses of THC, quite higher than the doses of THC used by cannabis abusers, the concentration of the steroid hormone pregnenolone increases in the brain. Pregnenolone then binds to a specific site on the CB1 receptors, distinct for the one of CB1 agonists and THC, and acts as an endogenous signaling specific inhibitor of the CB1 receptors. Pregnenolone cannot be used as a pharmacological treatment because it is poorly bioavailable, has a very short half-life and is converted downstream to active steroids. Aelis Farma, in collaboration with researchers from the Institut National de la Santé et de la Recherche Médicale (INSERM), has developed a new pharmacological class, the synthetic signaling specific inhibitor of the CB1 receptor (sCB1-SSi) AEF0117, by modifying pregnenolone's chemical structure to prevent conversion to active steroids, and to increase absorption and biological stability while maintaining THC antagonism.

To date, 3 clinical studies have been completed with AEF0117 including 2 phase 1 studies in healthy volunteers (AEF0117-101 single ascending dose study and AEF0117 102, multiple ascending dose study), and a phase 2a trial in cannabis users (AEF0117 201). The phase 1 studies showed good safety and tolerability of AEF0117 in the dose range tested (0.2 mg as single dose and 0.6-6 mg/day as single and multiple doses) and the phase 2a trial found that the 1 mg/day dose of AEF0117 significantly reduced both the abuse-related subjective effects of cannabis and its self-administration, while the 0.06 mg dose did not. Importantly, AEF0117 was well tolerated in daily cannabis smokers, with no evidence of precipitated withdrawal, physical, or psychological discomfort. There were no SAEs and a limited number of TEAEs. These results confirm preclinical data showing that AEF0117 does not function as an orthosteric antagonist and does not produce any of the adverse effects associated with rimonabant. Thus, AEF0117 is to our knowledge the first medication to safely and robustly attenuate the positive subjective and reinforcing effects of cannabis in participants with CUD.

In the 3 early studies conducted with AEF0117, AEF0117 was administered orally after a light breakfast. AEF0117 showed a good bioavailability and favorable, dose-proportional pharmacokinetics . In this protocol, the effects of food on AEF0117 bioavailability in healthy volunteers will be investigated by comparing the rate and extent of AEF0117 when 1 mg AEF0117 is administered in fed state versus fasting state.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date. This trial will provide data on the effect of food on the oral bioavailability of AEF0117 to support the next stage of the clinical development of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking male or female of any race, 18 to 55 years old, both inclusive.
2. Both males and female participants must use highly effective contraception during the entire trial period. Male participants should refrain from donating sperm or planning a pregnancy throughout the trial. Male participants must agree to use double-barrier contraceptive methods: male condoms and spermicide. FHeterosexually active females are only eligible if they are documented to be surgically sterile (e.g., hysterectomy, tubal ligation) or post-menopausal (amenorrhea >1 year and follicle-stimulating hormone [FSH] >25.8 mIU/mL) and with a negative pregnancy test.
3. Body mass index (BMI) of 22.0-35.0 kg/m2 (inclusive).
4. Be informed of the nature of the trial and provide signed informed consent to participate in the trial prior to any trial-specific procedures.
5. After being shown the high fat meal, understands and accepts that the entire meal should be consumed within 30 minutes.
6. Be legally competent and able to communicate effectively (in English) with trial personnel.

Exclusion Criteria:

1. Tobacco cigarette smokers within the last 3 months prior to dosing with trial drug.
2. Any disease or condition that might compromise the cardiovascular, hematologic, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer and cholecystectomy) systems, or any clinical laboratory values assessed as potentially clinically significant by the investigator .
3. Blood pressure outside normal range (140/80 mmHg systolic/diastolic) and considered potentially clinically significant.
4. Congenital long QT syndrome, history of prolonged QT in the 3 months prior to screening.
5. A corrected QT interval (Fridericia's - QTcF) >450 msec (male) or >470 msec (female) or history of risk factors for Torsades de Pointes.
6. A history of alcoholism or drug addiction within the past 2 years, recent use (in the last month) of any illicit drugs, or positive results from a urine screen for substances of abuse or from an alcohol breath test.
7. A history of or current serious mental illness including active or recent suicidal ideation, severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder) and/or an abnormal Columbia-Suicide Severity Rating Scale (C-SSRS) result.
8. Severe learning disability, brain damage, or pervasive developmental disorder.
9. A history of difficulty donating blood or inadequate venous access.
10. Clinically significant anemia or low hemoglobin (levels <9 g/dL) at screening, or donation of >250 mL of blood or plasma within the 30 days prior to prior to receiving trial drug or received any blood and plasma for medical/surgical reasons within the 30 days prior to prior to receiving trial drug, or intention to donate blood or plasma within 1 month after receiving trial drug.
11. History of or current HIV or hepatitis B or C.
12. History of COVID-19 within 4 weeks prior to Day -1, or positive COVID 19 test, according to standard procedures at the site, at screening or Day 1.
13. Positive serum pregnancy test (ß-hCG) at screening or positive urine pregnancy test at Day 1 confirmed by a serum pregnancy test result.
14. Allergies to the trial drug and known allergies to pregnenolone or to corn and corn derivatives.
15. Use of any prescription or over-the-counter drug therapy, including psychoactive and/or psychotropic medication, herbal, homeopathic, vitamins, minerals, and nutritional supplements, bodybuilding supplements unapproved by the sponsor, within 2 weeks prior to receiving the trial drug (for drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
16. Use of a drug therapy, or diet or supplements (e.g., St. John's Wort) food and fruit juices (e.g., grapefruit juice) known to induce or inhibit hepatic drug metabolism within 30 days prior to receiving trial drug or during the trial.
17. Legal status that would interfere with participation.
18. Unable to follow the restrictions outlined in the protocol.
19. Ingestion of an investigational drug or product, or participation in a drug trial within a period of 90 days prior to receiving trial drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, PhD, Principal Investigator — Substance Use Research Center
Locations (1):
- Substance Use Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AEF0117 1.0 mg in Fasted Condition: 11 participants receive 1 dose of AEF0117 1 mg in fasted condition
- AEF0117 1.0 mg in Fed Condition: 11 participants receive 1 dose of AEF0117 1 mg fed condition
Period: Overall Study
Arm/Group | AEF0117 1.0 mg in Fasted Condition | AEF0117 1.0 mg in Fed Condition
Started | 11 | 11
Completed | 11 | 7
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AEF0117 1.0 mg in Fasted Condition | AEF0117 1.0 mg in Fed Condition | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 85.45 (11.46) | 81.25 (13.65) | 83.35 (12.48)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.195 (3.161) | 26.307 (3.145) | 26.751 (3.110)

OUTCOME MEASURES:

1. Primary Outcome: Cmax of AEF0117
Description: Plasma concentration maximum(Cmax) of a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions.
Time Frame: up to 312 hours after dosing
Population: 1 subject in the Fed group was excluded from the pharcokinetic population due to missing data with 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- AEF0117 1.0 mg Once Daily (QD) in Fed Condition: 11 participants receive 1 dose of AEF0117 1 mg fed condition
Arm/Group | AEF0117 1.0 mg Once Daily (QD) in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
pg/mL | 6.87 (38.0) | 3.76 (28.6)
Statistical Analysis 1: Comparison: AEF0117 1.0 mg Once Daily (QD) in Fed Condition vs AEF0117 1.0 mg in Fasted Condition; Test type: Equivalence — Bioequivalence was declared if the 90% CI is included in between 0.8 and 1.25 range; p = 0.0079, t-test, 2 sided; Ratio of the geometric means = 1.824, 90% CI 2-sided [1.321 to 2.518]

2. Primary Outcome: Tmax of AEF0117
Description: Time to maximum plasma concentration (tmax) of a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions.
Time Frame: up to 312 hours after dosing
Population: 1 subject in the Fed group was excluded from the pharcokinetic population due to missing data with 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | AEF0117 1.0 mg Once Daily (QD) in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
hours | 3.5165 [2.0170 to 6.0000] | 3.0000 [2.0000 to 3.0000]

3. Primary Outcome: AUC (Area Under Curve) t to Last Concentration of AEF0117
Description: Area under the plasma concentration (AUC to Last Nonzero Conc) based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions
Time Frame: up to 312 hours after dosing
Population: 1 subject in the Fed group was excluded from the pharcokinetic population due to missing data with 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*pg/mL
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
hours*pg/mL | 61.50 (22.0) | 34.43 (27.8)
Statistical Analysis 1: Comparison: AEF0117 1.0 mg in Fed Condition vs AEF0117 1.0 mg in Fasted Condition; Test type: Equivalence — Bioequivalence was declared if the 90% CI is included in between 0.8 and 1.25 range; p < 0.0001, t-test, 2 sided; ratio of geometric means = 1.786, 90% CI 2-sided [1.470 to 2.170]

4. Secondary Outcome: Lowest Peak Plasma (Cmin) of AEF0117 Plasma Exposure
Description: Lowest Peak Plasma (Cmin) induced by a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions
Time Frame: up to 312 hours after dosing
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
pg/mL | 373.9108 (149.2681) | 154.1652 (62.7416)

5. Secondary Outcome: Terminal Elimination Half-life (t1/2) of AEF0117
Description: Terminal elimination half-life (t1/2) based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions
Time Frame: up to 312 hours after dosing
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
hours | 170.5580 [32.5230 to 212.9730] | 212.3460 [181.7600 to 242.7210]

6. Primary Outcome: AUC (Area Under Curve) t to Infinity Observed of AEF0117
Description: Area under the plasma concentration (AUC infinity obs) based on serial blood sample collections and plasma AEF0117 concentration after fed conditions relative to fasting conditions
Time Frame: up to 312 hours after dosing
Population: 1 subject in the Fed group was excluded from the pharcokinetic population due to missing data with 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*pg/mL
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
hours*pg/mL | 70.86 (23.7) | 42.14 (26.0)
Statistical Analysis 1: Comparison: AEF0117 1.0 mg in Fed Condition vs AEF0117 1.0 mg in Fasted Condition; Test type: Equivalence — Bioequivalence was declared if the 90% CI is included in between 0.8 and 1.25 range; p = 0.0002, t-test, 2 sided; ratio of geometric means = 1.681, 90% CI 2-sided [1.382 to 2.046]

7. Primary Outcome: Bioavailibility of AEF0117 (Tlag)
Description: Tlag is the Time point of first quantifiable concentration after dose administration
Time Frame: up to 312 hours after dosing
Population: 1 subject in the Fed group was excluded from the pharmacokinetic population due to missing data with 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 10 | 11
hours | 0.5000 [0.0000 to 1.0000] | 0.0000 [0.0000 to 0.0000]

8. Secondary Outcome: Incidence of Treatment-Emergent Adverse Event
Description: Number of participant reporting at least one Adverse Event
Time Frame: up to 312 hours after AEF0217 dosing
Measure: Count of Participants; unit: Participants
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
Number analyzed (Participants) | 11 | 11
Participants | 3 | 6

ADVERSE EVENTS:
Time Frame: from D1 (IP administration) until D14
Groups:
- AEF0117 1.0 mg in Fasted Condition: 11 participants receive 1 dose of AEF0117 1 mg fasted condition
Arm/Group | AEF0117 1.0 mg in Fed Condition | AEF0117 1.0 mg in Fasted Condition
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEF0117 1.0 mg in Fed Condition (N=11) | AEF0117 1.0 mg in Fasted Condition (N=11)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Brain Fog (Nervous system disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05451017/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT05451017/SAP_001.pdf